CLINICAL TRIAL: NCT01447160
Title: Effectiveness of Facet Joint Infiltration in Low Back Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Federal University os Sao Paulo, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUSao Paulo
Record Dates: First submitted 2011-07-29; First posted 2011-10-06 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-07

CONDITIONS: Low Back Pain
Keywords: facet joint; back pain; osteoarthritis; infiltration
MeSH Terms: conditions — Low Back Pain; Back Pain; Osteoarthritis | interventions — Cortisone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- facet joint infiltration (Experimental): The experimental group will be submitted to intra-articular infiltration of six facet joints (L3/L4;L4/L5;L5/S1 bilaterally) with triamcinolone hexacetonide
  Interventions: Drug: Cortisone
- intramuscular injection (Active Comparator): The control group which were submitted to triamcinolone acetonide intramuscular injection of six lumbar paravertebral points
  Interventions: Drug: Cortisone

INTERVENTIONS:
Drug: Cortisone — intraarticular infiltration with 1ml of triamcinolone hexacetonide versus intramuscular injection with 1 ml of triamcinolone acetonide

SUMMARY:
The purpose of this study is to evaluate the effectiveness of facet joint infiltration with corticosteroids in the treatment of low back pain due to facet joint osteoarthritis.

DETAILED DESCRIPTION:
Sixty subjects with diagnostic of facet joint syndrome will be enrolled in the study.

They were randomized into experimental and control groups. The experimental group will be submitted to intra-articular infiltration of six facet joints. The control group will be submitted to intramuscular injection of six lumbar paravertebral points. After the randomization, all subjects will be assessed by an investigator blinded to the groups. The assessment will be taken just before the interventions (T0) and them 7 , 30 , 90 and 180 days after the interventions. The following assessment instruments will be used: pain visual analogical scale (VAS) (0-10cm), pain visual analogical scale during extension of the spine (VAS E) (0-10cm), Likert scale for improving (0-5), percentage scale of subjective improving perception(0-100%), Rolland-Morris questionnaire (0-24), short health survey questionnaire (SF36), accountability of medications taken for back pain: analgesics and non-steroidal antiinflammatories (NSAIDs).

ELIGIBILITY:
Inclusion Criteria:

* low back pain up to 3 months
* pain on back extension
* radiologic findings of facet joint osteoarthritis

Exclusion Criteria:

* other causes of back pain
* fibromyalgia
* diabetes, arterial hypertension or glaucoma not well controlled
* patients with contrast allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
pain visual analogic scale | baseline
  pain visual scale graduated from zero to ten
pain visual analogic scale | 4 weeks
  pain visual analogic scale graduated 0--10
pain visual analogic scale | 12 weeks
  pain visual analogic scale graduated 0--10
pain visual analogic scale | 24 weeks
  pain visual analogic scale graduated 0--10

SECONDARY OUTCOMES:
Rolland Morris questionnaire | baseline
  assess functional capacity
Rolland Morris questionnaire | 4 weeks
  assess functional capacity
Rolland Morris questionnaire | 12 weeks
  assess functional capacity
Rolland Morris questionnaire | 24 weeks
  assess functional capacity
SF-36 questionnaire | baseline
  assess quality of life
SF-36 questionnaire | 4 weeks
  assess quality of life
SF-36 questionnaire | 12 weeks
  assess quality of life
SF-36 questionnaire | 24 weeks
  assess quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Luiza Ribeiro, doctor, Principal Investigator — Sao Paulo Federal University
Locations (1):
- Sao Paulo federal University, São Paulo, São Paulo, Brazil